CLINICAL TRIAL: NCT01753518
Title: A Randomized Clinical Trial of Subcuticular Staples Versus Subcuticular Suture for Cesarean Section Skin Closure
Brief Title: A Clinical Trial of Subcuticular Staples Versus Subcuticular Suture for Cesarean Section Skin Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Margaret L. Dow, M.D. (Other)
Responsible Party: Sponsor-Investigator, Margaret L. Dow, M.D., M.D., Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-003183
Record Dates: First submitted 2012-12-05; First posted 2012-12-20 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Surgical Wound
Keywords: Subcuticular suture; Subcuticular staple; Skin closure; Incision closure; Wound
MeSH Terms: conditions — Surgical Wound; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcuticular suture (Active Comparator): Subcuticular suture has been used for many years to close skin incisions.
  Interventions: Device: Subcuticular suture
- Subcuticular staple (Active Comparator): Subcuticular staples are a newer modality than suture, but are currently an accepted and widely used skin closure technique.
  Interventions: Device: Subcuticular staple

INTERVENTIONS:
Device: Subcuticular suture — subcuticular Monocryl suture closure
  Other Names: Monocryl
  Arms: Subcuticular suture
Device: Subcuticular staple — subcuticular staple wound closure with INSORB 20 device
  Other Names: Insorb
  Arms: Subcuticular staple

SUMMARY:
Currently, the way doctors close the skin during cesarean section is different between surgeons and there is little evidence to support the use of one kind of closure over the other. At the Mayo Clinic Family Birth Center, skin is currently closed using an absorbable suture (or stitch), placed within the top layer of skin. At other institutions, a metal staple is often used to close the skin.

There is a new technique that uses special absorbable staples just beneath the skin. This technology may be equal to, or possibly better than, current skin closure techniques. However, there is currently little data to show how it compares. The purpose of this study is to compare the absorbable staple to the currently used absorbable suture. The data from this study will then be used to help determine the best technique for skin closure.

DETAILED DESCRIPTION:
Cesarean section is one of the most frequently performed surgical procedures worldwide. In the United States, the proportion of deliveries by cesarean has increased from approximately 21% in 1996 to 32.8% in 2010. Ultimately, the rising incidence of cesarean delivery results in increased surgical morbidity; including pain, blood loss, and surgical site infections, which leads to an increase in overall hospitalization days and healthcare costs. This volume of surgical procedures also carries the risk of blood and body fluid exposures to surgical staff. Suture needles contribute to 43.4% of all sharps injuries in surgical settings and 51.5% of sharp injuries to surgeons alone. Additionally, it was discovered that 20% of blood borne pathogen exposures on the Mayo Clinic Rochester campus in 2011 occurred in the Department of Obstetrics and Gynecology. Therefore, any quality improvement measure regarding cesarean sections has the potential to significantly impact overall surgical morbidity, bloodborne pathogen exposure, and healthcare costs at our institution. Reviews of current literature show a lack of evidence for many of the surgical steps during cesarean procedures. Thus, there is an urgent need to define evidence-based surgical techniques for each step, from incision to closure.

The optimal skin closure technique is simple, quick, cost-effective, and provides adequate tissue approximation with a good cosmetic outcome while minimizing the risk of infection, dehiscence, and pain. Ideally, needlestick injuries would also be eliminated. It is currently unknown which skin closure method is superior with regard to these outcomes.

The INSORB 20 (Incisive Surgical) is a new, single-use device for skin closure that aims to combine the speed of a staple with the cosmetic outcome of a subcuticular suture, while eliminating the need for staple removal. Additionally, it should reduce the incidence of needlestick injury. INSORB also claims to result in a "low maintenance wound" with less surgical site infection, lower inflammation, and increased patient comfort and satisfaction. However, data is limited comparing INSORB to the current standards of care (either staples or suture).

The purpose of this study is to determine if the new absorbable subcuticular staples (INSORB) improves outcomes compared to the current standard absorbable subcuticular suture for skin closure in cesarean sections.

ELIGIBILITY:
Inclusion criteria:

* Gestational age ≥ 24 weeks
* Scheduled cesarean section for any indication
* Pfannenstiel incision
* Singleton gestation

Exclusion criteria:

* Failure to consent
* Gestational age < 24 weeks
* Vaginal delivery
* Intrauterine fetal death
* Multifetal gestation
* Suspected infection, i.e. chorioamnionitis
* BMI > 50

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tessmer-Tuck, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Tuuli MG, Rampersad RM, Carbone JF, Stamilio D, Macones GA, Odibo AO. Staples compared with subcuticular suture for skin closure after cesarean delivery: a systematic review and meta-analysis. Obstet Gynecol. 2011 Mar;117(3):682-690. doi: 10.1097/AOG.0b013e31820ad61e. PMID 21343772
- [Background] Jagger J, Bentley M, Tereskerz P. A study of patterns and prevention of blood exposures in OR personnel. AORN J. 1998 May;67(5):979-81, 983-4, 986-7 passim. doi: 10.1016/s0001-2092(06)62623-9. PMID 9592605
- [Background] Jenkins TR. It's time to challenge surgical dogma with evidence-based data. Am J Obstet Gynecol. 2003 Aug;189(2):423-7. doi: 10.1067/s0002-9378(03)00587-8. PMID 14520211
- [Background] Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery. Am J Obstet Gynecol. 2005 Nov;193(5):1607-17. doi: 10.1016/j.ajog.2005.03.063. PMID 16260200
- [Background] Walsh CA. Evidence-based cesarean technique. Curr Opin Obstet Gynecol. 2010 Apr;22(2):110-5. doi: 10.1097/GCO.0b013e3283372327. PMID 20216417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic Family Birth Center (labor and delivery) in Rochester, Minnesota. Subjects were recruited from December 2012 until the end of April 2014.
Pre-assignment Details: 220 subjects were randomized to suture or absorbable subcuticular staples and 206 were included in the final analysis with 103 in each group. One subject crossed over from absorbable subcuticular staples to suture intraoperatively, because the attending surgeon was not comfortable with the staple closure device.
Period: Intention-to-Treat Analysis
Arm/Group | Subcuticular Suture | Subcuticular Staple
Started | 110 | 110
Completed | 103 | 103
Not Completed | 7 | 7
Not completed — Missing consent form | 5 | 3
Not completed — Multifetal gestation | 2 | 3
Not completed — Body Mass Index>50 | 0 | 1
Period: Postpartum Follow-up
Arm/Group | Subcuticular Suture | Subcuticular Staple
Started | 103 | 103
Completed | 81 | 88
Not Completed | 22 | 15
Not completed — Lost to Follow-up | 22 | 15

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat Analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcuticular Suture | Subcuticular Staple | Total
Number analyzed (Participants) | 103 | 103 | 206
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [27 to 33] | 31 [27 to 34] | 30.5 [27 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 103 | 206
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 103 | 103 | 206
Resident year of postgraduate education [Median (Inter-Quartile Range); unit: years] | 2 [2 to 4] | 2 [2 to 3] | 2 [2 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Total Surgical Time, All Resident Levels
Description: Total surgical time was defined as the time from incision start to incision completion. Measured for all resident education levels (1 to 4 years postgraduate).
Time Frame: Measured at the time of the procedure (day 1), approximately 1 hour after incision start
Population: Intention-to-Treat
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 103 | 103
minutes | 58.0 [50.4 to 68.2] | 54.0 [44.9 to 63.6]
Statistical Analysis 1: Comparison: Subcuticular Suture vs Subcuticular Staple; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Total Number of Participants With Postoperative Complications
Description: Postoperative complications were assessed by chart review.
Time Frame: From the day of the procedure (Day 1) for 6 weeks
Population: The number of participants analyzed was reduced because some patients did not return for postpartum followup visits.
Measure: Number; unit: participants
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 93 | 96
participants | 7 | 6
Statistical Analysis 1: Comparison: Subcuticular Suture vs Subcuticular Staple; Test type: Superiority or Other; p = 0.73, Chi-squared

3. Secondary Outcome: Participants With Postoperative Complications, by Type
Description: Postoperative complications were assessed by chart review.
Time Frame: From the day of the procedure (Day 1) for 6 weeks
Population: Participants could have experienced more than one type of postoperative complication. Note: wound dehiscence is a surgical complication in which a wound ruptures along surgical suture. A seroma is a pocket of clear serous fluid. A hematoma is a localized swelling that is filled with blood caused by a break in the wall of a blood vessel.
Measure: Number; unit: participants
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 93 | 96
participants
  Staple Expulsion or Suture Trimming | 0 | 3
  Surgical Site Infection | 4 | 1
  Superficial Wound Separation | 4 | 1
  Complete Wound Dehiscence | 0 | 0
  Seroma | 1 | 0
  Hematoma | 0 | 2
  No Postoperative Complications | 86 | 90
Statistical Analysis 1: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison for staple expulsion or suture trimming; Test type: Superiority or Other; p = 0.25, Fisher Exact
Statistical Analysis 2: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison for Surgical Site Infection; Test type: Superiority or Other; p = 0.06, Fisher Exact
Statistical Analysis 3: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison for Superficial Wound Separation; Test type: Superiority or Other; p = 0.21, Fisher Exact
Statistical Analysis 4: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison for Seroma; Test type: Superiority or Other; p = 0.49, Fisher Exact
Statistical Analysis 5: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison for Hematoma; Test type: Superiority or Other; p = 0.50, Fisher Exact

4. Secondary Outcome: Postoperative Pain
Description: Post-operative pain was assessed by pain medication use through chart review.
Time Frame: From day of procedure until end of hospital stay (typical dismissal on day 4)
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 103 | 103
mg
  Tylenol | 12000 [11000 to 13000] | 12000 [9000 to 13000]
  Ibuprofen | 5400 [3600 to 6000] | 4800 [3600 to 6000]
  Toradol | 45 [45 to 45] | 45 [45 to 45]
  Oxycodone | 60 [30 to 100] | 60 [25 to 100]
Statistical Analysis 1: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between the arms for Tylenol use; Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between the arms for Ibuprofen use; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between the arms for Toradol use; Test type: Superiority or Other; p = 0.85, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between the arms for Oxycodone use; Test type: Superiority or Other; p = 0.78, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Subjects Requiring Patient-controlled, Alternative Oral, or Single Dose IV/IM Analgesic
Description: Post-operative pain was assessed by pain medication use through chart review. These subjects required patient-controlled analgesia, or alternative oral analgesic, or a single dose of intravenous (IV) or intramuscular (IM) analgesic. Alternative oral analgesics included hydromorphone, hydrocodone/acetaminophen, or oxycodone/acetaminophen .
Time Frame: From day of procedure until end of hospital stay (typical dismissal on day 4)
Measure: Number; unit: participants
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 97 | 99
participants
  Patient-controlled analgesia | 5 | 6
  Alternative oral analgesic | 6 | 9
  Single dose IV/IM analgesic | 16 | 22

6. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction was measured by questionnaire at the time of dismissal from the hospital and at their 6 week postpartum/postoperative exam. There were 4 questions: How satisfied are you with the appearance of your skin incision? How willing are you to recommend this same skin closure to a friend? How willing are you to have this same skin closure for your next cesarean section? What is your overall satisfaction with your surgical procedure, including the skin incision? For reporting purposes, possible answers for each item were grouped into negative (not at all, not very, or no opinion), or positive (somewhat or extremely).
Time Frame: At the time of dismissal (typically day 3 or 4) and at 6 weeks postoperative appointment
Population: The reduction in the number of participants analyzed is due to not all participants completing the questionnaire, and all the questions. For appearance of incision, N=58:69. For willingness to use treatment again, N=59:68.
Measure: Number; unit: participants
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 59 | 69
participants
  Appearance of incision: negative | 3 | 6
  Appearance of incision: positive | 55 | 63
  Would recommend: negative | 11 | 6
  Would recommend: positive | 48 | 63
  Willingness (again): negative | 8 | 7
  Willingness (again): positive | 51 | 61
  Overall satisfaction: negative | 4 | 2
  Overall satisfaction: positive | 55 | 67
Statistical Analysis 1: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison for negative responses to "Appearance of incision" question; Test type: Superiority or Other; p = 0.51, Fisher Exact
Statistical Analysis 2: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison for negative responses to "Would recommend treatment to friends" question; Test type: Superiority or Other; p = 0.098, Chi-squared
Statistical Analysis 3: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison of negative responses to "Willingness to use treatment again" question; Test type: Superiority or Other; p = 0.57, Chi-squared
Statistical Analysis 4: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison of negative responses to "Overall satisfaction" question; Test type: Superiority or Other; p = 0.41, Fisher Exact

7. Secondary Outcome: Surgeon Satisfaction (Per Procedure)
Description: Surgeon satisfaction was assessed by a 3-question questionnaire immediately after performing the procedure. The questions were: How satisfied are you with the appearance of the skin incision?" "How willing are you to recommend this skin closure (whether it was staples or suture) to a patient?" "How willing are you to use this skin closure (whether it was staples or suture) for your next cesarean section?" There were 5 possible responses to each question (not at all, not very, no opinion, somewhat, extremely), with "not at all,' "not very," and "no opinion" being a negative response, and "somewhat" and "extremely " being a positive response. Categories reported were negative, (including no opinion), and positive.
Time Frame: Immediately after the procedure (day 1)
Population: A satisfaction survey wasn't completed for all of the procedures (103 per arm), so the reporting population is 91 for the suture arm, and 96 for the staple arm.
Measure: Number; unit: Surgeons reporting per category
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 91 | 96
Surgeons reporting per category
  Appearance of incision: negativ | 6 | 7
  Appearance of incision: positive | 85 | 89
  Recommend: negative | 14 | 3
  Recommend: positive | 77 | 93
  Willingness to use again: negative | 16 | 2
  Willingness to use again: positive | 75 | 94
Statistical Analysis 1: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for "appearance of incision."; Test type: Superiority or Other; p = 0.85, Chi-squared
Statistical Analysis 2: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for "recommend treatment."; Test type: Superiority or Other; p = 0.004, Chi-squared
Statistical Analysis 3: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for "willingness to use treatment again."; Test type: Superiority or Other; p < 0.001, Chi-squared

8. Primary Outcome: Skin Closure Time, All Resident Levels
Description: Measured for all resident education levels (1 to 4 years postgraduate).
Time Frame: Measured at the time of the procedure (day 1), approximately 1 hour after incision start
Population: Intention-to-Treat
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 103 | 103
minutes | 8.5 [6.2 to 10.5] | 2.6 [1.8 to 4.0]
Statistical Analysis 1: Comparison: Subcuticular Suture vs Subcuticular Staple; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Cosmetic Outcome
Description: The cosmetic outcome will be assessed by patients and a blinded observer at the 6 week postpartum/postoperative exam using the Patient Observer Scar Assessment Scale (POSAS). The POSAS consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically. Each item of both scales has a 10-point score, with 10 indicating the worst imaginable scar or sensation. The lowest score is '1', and corresponds to the situation of normal skin (normal pigmentation, no itching etc), and goes up to the worst imaginable. Besides the six items the 'Overall Opinion' of the scar quality is scored separately of both patients and observers. Again, a 10-point scale is used in which 10 corresponds to the worst imaginable scar.
Time Frame: Measured at 6 week postoperative appointment
Population: Not all patients or observers completed the scales. For the six items on the patient scale, N=44:52, but the overall opinion responding was N=43:51. For the observer scale the number responding was N=43:52 for vascularity, thickness, pliability, and surface area. N=42:52 for pigmentation and relief; N=42:50 for overall opinion.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Subcuticular Suture | Subcuticular Staple
Number analyzed (Participants) | 44 | 52
units on a scale
  Patient: scar painful | 2.2 [1 to 3] | 1.8 [1 to 2]
  Patient: scar itching | 2.2 [1 to 3] | 1.9 [1 to 3]
  Patient: scar color is different | 5.3 [2 to 8] | 3.9 [1.5 to 6]
  Patient: scar stiffness is different | 5.0 [2 to 8] | 3.7 [2 to 6]
  Patient: scar thickness is different | 4.6 [2 to 7.5] | 4.0 [1.5 to 6.5]
  Patient: scar more irregular | 4.4 [2 to 6] | 3.6 [1 to 5.5]
  Patient: scar overall opinion | 4.4 [3 to 6] | 3.8 [2 to 5]
  Observer: vascularity | 2.9 [2 to 4] | 2.8 [2 to 3]
  Observer: pigmentation | 3.2 [2 to 4] | 2.5 [2 to 3]
  Observer: thickness | 2.7 [2 to 3] | 2.6 [2 to 3]
  Observer: relief | 2.5 [1 to 3] | 2.6 [2 to 3]
  Observer: pliability | 2.7 [1 to 4] | 2.8 [2 to 3]
  Observer: surface area | 2.5 [2 to 3] | 2.5 [2 to 3]
  Observer: overall opinion | 2.8 [2 to 3] | 2.6 [2 to 3]
Statistical Analysis 1: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for patient: scar painful; Test type: Superiority or Other; p = 0.35, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for patient: scar itching; Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for patient: scar color is different; Test type: Superiority or Other; p = 0.034, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for patient: scar stiffness is different; Test type: Superiority or Other; p = 0.041, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for patient: scar thickness is different; Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for patient: scar more irregular; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for patient: overall opinion; Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for observer: vascularity; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for observer: pigmentation; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for observer: thickness; Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for observer: relief; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for observer: pliability; Test type: Superiority or Other; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for observer: surface area; Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Subcuticular Suture vs Subcuticular Staple; Comparison between arms for observer: overall opinion; Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Post operative complications were collected from December 2012 through June 2014.
Description: Not all subjects returned for their postpartum appointment, so the reporting population is Suture (N=93) and Staples (N=96). Subjects could have experienced more than one category of complications.
Arm/Group | Subcuticular Suture | Subcuticular Staple
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/96
Other Adverse Events (participants affected / at risk) | 7/93 | 6/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcuticular Suture (N=93) | Subcuticular Staple (N=96)
Staple expulsion or suture trimming (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3)
Surgical Site Infection (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0)
Superficial Wound Separation (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
Seroma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — A seroma is a pocket of clear serous fluid that sometimes develops in the body after surgery.
Hematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) — A hematoma is a circumscribed collection of blood, usually clotted, in a tissue or organ, caused by a break in a blood vessel.

LIMITATIONS AND CAVEATS:
The data are limited by the lack of diversity, and there may be racial or genetic differences in wound healing confounding the results. This trial was not powered for postoperative wound complications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes